CLINICAL TRIAL: NCT01498809
Title: Neural and Mechanical Baroreflex Sensitivity and Cerebral Blood Flow
Brief Title: Blood Pressure and Brain Blood Flow Regulation After Midodrine Administration in Those With Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Other Study IDs: H11-02823
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Orthostatic Intolerance
Keywords: Orthostatic intolerance in people with spinal cord injury
MeSH Terms: conditions — Orthostatic Intolerance | interventions — Midodrine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Midodrine — Single 10 mg dose
  Other Names: Amatine, ProAmatine, Gutron

SUMMARY:
This project aims to evaluate the physiological effects of Midodrine administration during orthostatic challenge in those with high level spinal cord injury. Midodrine has been shown to improve orthostatic symptoms in those with spinal cord injury but the physiological mechanisms influenced have not been identified. The investigators will examine key physiological components influencing orthostatic tolerance. The investigators will do this, by measuring the baroreflex, and brain blood flow autoregulation (the ability to maintain brain blood flow) before during and after the sit-up test. Two sit-up tests will occur; one before Midodrine administration, and one after administration of a 10mg dose of Midodrine.

ELIGIBILITY:
Inclusion Criteria:

* To be included in the study, participants must have sustained a traumatic spinal cord injury within the ages of 18-49 years.
* Also, participants must have an injury level above the 6th thoracic vertebrae and be a non-smoker for a minimum of one year.

Exclusion Criteria:

* Any participants with a history of cardiovascular disease, pulmonary disease or diabetes mellitus will not be eligible.
* Also, participants will not be eligible to take part in study if they experiences acute distress, or are taking medications known to influence cardiovascular function.
* Patient will be not eligible for the study if he/she has known adverse reaction to Midodrine.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals with spinal cord injury currently in primary care (less than one year post injury)
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Baroreflex sensitivity | Immediately after drug administration (30 mins)

SECONDARY OUTCOMES:
Cerebral autoregulation | Thirty minutes after administration

CONTACTS AND LOCATIONS:
Overall Officials: Darren Warburton, PhD, Principal Investigator — University of British Columbia; Andrei Krassioukov, MD PhD, Principal Investigator — GF Strong Hospital University of British Columbia
Locations (1):
- GF Strong Hospital and Rehabilitation Centre, Vancouver, British Columbia, Canada